CLINICAL TRIAL: NCT02088684
Title: A Phase Ib/II Study of LEE011 in Combination With Fulvestrant and BYL719 or BKM120 in the Treatment of Postmenopausal Women With Hormone Receptor Positive, HER2 Negative Locally Recurrent or Advanced Metastatic Breast Cancer
Brief Title: Study of LEE011 With Fulvestrant and BYL719 or BKM120 in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011X2108
Record Dates: First submitted 2014-03-12; First posted 2014-03-17 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Hormone receptor positive, HER2 negative
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Alpelisib; Fulvestrant; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LEE011 + BKM120 + fulvestrant (Experimental): LEE011 - 28 day cycles (21 days followed by a 7 day break - dose escalating) BKM120 - daily (dose escalating) fulvestrant - i.m. - 500 mg given on day 1 and day 15 of Cycle 1, then on Day 1 of each subsequent cycle.
  Interventions: Drug: LEE011; Drug: fulvestrant; Drug: BKM120
- LEE011 + BYL719 + fulvestrant (Experimental): LEE011 - 28 day cycles (21 days followed by a 7 day break - dose escalating) BYL719 - daily (dose escalating) fulvestrant - i.m. - 500 mg given on day 1 and day 15 of Cycle 1, then on Day 1 of each subsequent cycle.
  Interventions: Drug: LEE011; Drug: BYL719; Drug: fulvestrant
- LEE011 + fulvestrant (Experimental): LEE011 - 28 day cycles (3 weeks on, 1 week off) or (continuous daily dosing - dose escalating) fulvestrant - 500 mg i.m. given on Day 1 and Day 15 of Cycle 1, then on Day 1 of each subsequent cycle.
  Interventions: Drug: LEE011; Drug: fulvestrant

INTERVENTIONS:
Drug: LEE011 — LEE011: supplied as capsules of dosage strength of 50 mg or 200 mg. The capsules will be differentiated through different sizes
Drug: BYL719 — BYL719: supplied as tablets of dosage strength of 10 mg, 50 mg or 200 mg. Tablets will be differentiated through different sizes and/or colors.
  Arms: LEE011 + BYL719 + fulvestrant
Drug: fulvestrant — Fulvestrant will be supplied according to local practice and regulation. Fulvestrant is a commercially available product, comes in 500 mg dose and is an injection for intramuscular (i.m.) administration.
Drug: BKM120 — BKM120: supplied as 10 mg or 50 mg capsules. The capsules will be differentiated through different sizes.
  Arms: LEE011 + BKM120 + fulvestrant

SUMMARY:
The purpose of this trial is to explore the clinical utility of the three investigational agents in HR+, HER2- breast cancer. LEE011 (CDK4/6 inhibitor), BKM120 (PI3K-pan class I-inhibitor) and BYL719 (PI3K-alpha specific class I inhibitor) in combination with fulvestrant.

This is a multi-center, open-label Phase Ib/II study. The Phase Ib portion of the study is a dose escalation to estimate the MTD and/or RP2D for three regimens: LEE011 with fulvestrant; LEE011 and BKM120 with fulvestrant; LEE011and BYL719 with fulvestrant.

The Phase II portion of the study was planned to be a randomized study to assess the anti-tumor activity as well as safety and tolerability of LEE011 with fulvestrant to LEE011 and BKM120 with fulvestrant, and LEE011 and BYL719 with fulvestrant in patients with ER+/HER2- locally advanced or metastatic breast cancer.

Approximately 216 adult women with ER+/HER2- locally advanced or metastatic breast cancer were planned to be enrolled.

DETAILED DESCRIPTION:
On 31-May-2016 Novartis's made the decision decision to not open the Phase II portion of the study, for business reasons. Sufficient data had already been collected and no additional data for the triplet combinations was needed. As a result, the Phase II portion of the trial was not opened.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, Hormone receptor positive (HR+), HER2 negative breast cancer
* Unlimited number of lines of endocrine therapy and up to two lines of cytotoxic chemotherapy in the metastatic setting (Phase Ib)
* Unlimited number of lines of endocrine therapy and one line of cytotoxic chemotherapy in the metastatic setting (Phase II)

Exclusion Criteria:

* HER2-overexpression in the patient's tumor tissue
* Inadequate bone marrow function or evidence of end-organ damage
* Severe or uncontrolled medical issues
* Diabetes mellitus

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2018-04-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities (DLTs) - Phase lb only | 28 days
  Dose limiting toxicities
Progression free survival (PFS) - Phase ll only | 36 months
  Progression Free Survival per RECIST v 1.1 by local investigator assessment

SECONDARY OUTCOMES:
Safety and Tolerability of the combinations of LEE011 with fulvestrant, LEE011 + BKM120 with fulvestrant and LEE011 + BYL719 with fulvestrant | 36 months
  Adverse Events (AEs), serious AEs (SAEs), changes in hematology and chemistry values, vital signs, electrocardiograms (ECGs), dose interruptions, reductions and dose intensity
Plasma concentration-time profiles of LEE011, BKM120, BYL719 and fulvestrant. | 36 months
  To characterize the PK profiles of LEE011, BKM120, BYL719, and fulvestrant when used in combination as well as to evaluate any other clinically significant metabolites that may be identified. PK parameters for LEE011, BKM120 and BYL719, including but not limited to Cmax, Cmin, Tmax, AUCtau, accumulation ratio (Racc),and Ctrough values for fulvestrant.
Overall Response Rate (ORR) | 36 months
  ORR is defined as the proportion of patients with a best overall response of complete response or partial response.
Duration of Response (DOR) | 36 months
  Duration of Response is calculated as the time from the date of first documented response (complete response (CR) or partial response (PR)) to the first documented date of progression or death due to underlying cancer.
Progression Free Survival (PFS) (phase l only) | 36 months
  PFS is the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.
Overall Survival (OS) - Phase II only | 36 months
  OS is defined as the time from date of randomization/start of treatment to date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last known date patient alive.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (3):
  - University of Alabama at Birmingham/ Kirklin Clinic Dept Onc, Birmingham, Alabama
  - Dana Farber Cancer Institute Onc. Dept., Boston, Massachusetts
  - Sarah Cannon Research Institute Onc Dept, Nashville, Tennessee
- Novartis Investigative Site, Lyon, France
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Madrid, Spain
- Novartis Investigative Site, Taipei, Taiwan ROC, Taiwan
- Novartis Investigative Site, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Tolaney SM, Im YH, Calvo E, Lu YS, Hamilton E, Forero-Torres A, Bachelot T, Maur M, Fasolo A, Tiedt R, Nardi L, Stammberger U, Abdelhady AM, Ruan S, Lee SC. Phase Ib Study of Ribociclib plus Fulvestrant and Ribociclib plus Fulvestrant plus PI3K Inhibitor (Alpelisib or Buparlisib) for HR+ Advanced Breast Cancer. Clin Cancer Res. 2021 Jan 15;27(2):418-428. doi: 10.1158/1078-0432.CCR-20-0645. Epub 2020 Sep 4. PMID 32887722
- See also: link to Novartis Clinical Trial result Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17409